CLINICAL TRIAL: NCT02782169
Title: Prophylactic Pregabalin to Decrease Pain During Medical Abortion: a Randomized Controlled Trial
Brief Title: Prophylactic Pregabalin to Decrease Pain During Medical Abortion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Hawaii (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SFPRF15-12
Record Dates: First submitted 2015-11-30; First posted 2016-05-25 (Estimated); Results first posted 2018-04-19 (Actual); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pregabalin (Active Comparator)
  Interventions: Drug: Pregabalin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pregabalin — Pregabalin 300 mg capsule (over encapsulated to maintain blinding)
  Arms: Pregabalin
Drug: Placebo — Matching placebo capsule with excipient to match Pregabalin
  Arms: Placebo

SUMMARY:
Medical abortion has been associated with significant pain. The objective of this trial is to determine whether one dose of pregabalin 300 mg, given during medical abortion in addition to the standard of care analgesics, will decrease experienced pain. Investigators will perform a randomized, double-blinded, placebo-controlled trial. Participant pain levels and side effects will be assessed at multiple time points, along with a measure of satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Requested and consented for pregnancy termination by medical abortion
* Willing and able to complete multiple electronic surveys

Exclusion Criteria:

* Previous participation in this trial
* Current use of pregabalin or gabapentin
* Contraindication to medical abortion with mifepristone and misoprostol
* Contraindication or allergy to ibuprofen, oxycodone, acetaminophen, or pregabalin
* Unable to understand and sign written informed consents in English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Women's Options Center, Honolulu, Hawaii, United States

REFERENCES:
- [Derived] Reynolds-Wright JJ, Woldetsadik MA, Morroni C, Cameron S. Pain management for medical abortion before 14 weeks' gestation. Cochrane Database Syst Rev. 2022 May 13;5(5):CD013525. doi: 10.1002/14651858.CD013525.pub2. PMID 35553047
- [Derived] Friedlander EB, Soon R, Salcedo J, Davis J, Tschann M, Kaneshiro B. Prophylactic Pregabalin to Decrease Pain During Medication Abortion: A Randomized Controlled Trial. Obstet Gynecol. 2018 Sep;132(3):612-618. doi: 10.1097/AOG.0000000000002787. PMID 30095762

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pregabalin | Placebo
Started | 56 | 54
Completed | 55 | 52
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pregabalin | Placebo | Total
Number analyzed (Participants) | 55 | 52 | 107
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.25 (5.45) | 27.19 (6.02) | 27.22 (5.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 52 | 107
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 18 | 12 | 30
  Native Hawaiian or Other Pacific Islander | 5 | 6 | 11
  Black or African American | 1 | 2 | 3
  White | 6 | 8 | 14
  More than one race | 23 | 21 | 44
  Unknown or Not Reported | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Maximum Pain Score Over Study Period
Description: reported on an 11-point numerical rating scale (NRS 0-10) where 0 indicates no pain and 10 indicates the most severe pain
Time Frame: Over 72 hours (measured at 0, 2, 6, 12, 24, and 72 hours)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 55 | 52
units on a scale | 5.0 (2.6) | 5.5 (2.2)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority; p = 0.32, t-test, 2 sided

2. Secondary Outcome: Number of Ibuprofen 800mg Tablets Used
Description: summed number of tablets used by each participant over the 72 hour study period
Time Frame: Over 72 hours (measured at 0, 2, 6, 12, 24, and 72 hours)
Measure: Median (Inter-Quartile Range); unit: tablets
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 55 | 52
tablets | 1 [0 to 4] | 2 [1 to 3]

3. Secondary Outcome: Number of Oxycodone/Acetominophen Tablets (5/325mg) Used
Description: summed number of tablets used by each participant over the 72 hour study period
Time Frame: Over 72 hours (measured at 0, 2, 6, 12, 24, and 72 hours)
Measure: Median (Inter-Quartile Range); unit: tablets
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 55 | 52
tablets | 0 [0 to 1] | 0.5 [0 to 1]

4. Secondary Outcome: Number of Participants Ever Experiencing Different Symptoms During Abortion
Description: A participant was included once if they ever reported a symptom during the 72 hour study period, not reflective of how long the symptom lasted. These were all commonly reported side effects during previous research on medication abortions and commonly reported side effects of pregabalin, so they were not included as adverse events.
Time Frame: Over 72 hours (measured at 0, 2, 6, 12, 24, and 72 hours)
Measure: Number; unit: participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 55 | 52
participants
  Nausea | 43 | 42
  Vomiting | 28 | 30
  Sleepiness | 47 | 39
  Dizziness | 45 | 26
  Headache | 28 | 17
  Blurred Vision | 15 | 7
  Diarrhea | 28 | 29
  Constipation | 6 | 15
  Dry Mouth | 22 | 25

5. Secondary Outcome: Satisfaction With Analgesia
Description: 5-point Likert scale (1=very dissatisfied, 2=dissatisfied, 3=neutral, 4=satisfied, 5=very satisfied)
Time Frame: Asked at time point of 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 55 | 52
Participants
  Very dissatisfied | 2 | 3
  Dissatisfied | 3 | 0
  Neutral | 12 | 13
  Satisfied | 11 | 24
  Very satisfied | 25 | 11
  No response | 2 | 1

ADVERSE EVENTS:
Arm/Group | Pregabalin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/52
Other Adverse Events (participants affected / at risk) | 0/55 | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No